CLINICAL TRIAL: NCT00911378
Title: A Randomized Controlled Trial on Weaning by Pressure Support Reduction Versus Spontaneous Breathing Trials in a Respiratory ICU
Brief Title: Pressure Support Reduction Versus Spontaneous Breathing Trials in Weaning From Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Dr. Ritesh Agarwal, Postgraduate Institute of Medical Education and Research
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: weaning2009
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Respiration, Artificial; Ventilator Weaning
Keywords: weaning; mechanical ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pressure support ventilation (Active Comparator): Patients in this arm are weaned by gradual reduction of pressure support
  Interventions: Procedure: Pressure support ventilation
- Spontaneous breathing trials (Active Comparator): Patients in this arm are weaned by T piece trials
  Interventions: Procedure: Spontaneous breathing trials

INTERVENTIONS:
Procedure: Pressure support ventilation — These patients are weaned by gradual reduction of pressure support and extubated when they tolerate a pressure support of 7 cm of water for one hour.
  Other Names: weaning by reduction of pressure support
  Arms: Pressure support ventilation
Procedure: Spontaneous breathing trials — These patients are weaned by giving a T piece trial with 8 cm of water pressure support and extubated when they tolerate it for one hour.
  Other Names: Weaning by T-piece trials
  Arms: Spontaneous breathing trials

SUMMARY:
This study is a comparison of two most commonly used modes of weaning and the outcomes in the two groups.

DETAILED DESCRIPTION:
Patients ventilated for more than 24 hours are randomized into two groups - one group of patients undergo gradual reduction of pressure support and in the other, T tube trials are used for weaning. The outcomes are compared in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients for more than 24 hours
* Satisfies weaning criteria
* RSBI < 80
* Ratio of PaO2/FiO2 > 250
* Arterial partial pressure of oxygen more than 60 mm Hg and carbon dioxide less than 50 mm Hg

Exclusion Criteria:

* Systolic blood pressure of less than 100
* Arterial partial pressure of oxygen less than 60 mm Hg
* Poor sensorium

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Rate of weaning failure | 48 hours from extubation

SECONDARY OUTCOMES:
Occurence of ventilator associated pneumonia | Until the date of discharge from hospital
Reintubation rates | 48 hours
Mortality rates | Until the time of discharge from hospital
Duration from start of weaning to extubation | In hospital stay
Role of various factors that may influence the weaning outcome and hence predict the probability of successful weaning in a patient | during ICU stay
The influence of weaning outcome on mortality and the other complications of mechanical ventilation | during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ashutosh Aggarwal, MD, DM, Study Director — Department of Pulmonary Medicine and Critical Care, Postgraduate Institute of Medical Education and Research
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

REFERENCES:
- [Result] Esteban A, Frutos F, Tobin MJ, Alia I, Solsona JF, Valverdu I, Fernandez R, de la Cal MA, Benito S, Tomas R, et al. A comparison of four methods of weaning patients from mechanical ventilation. Spanish Lung Failure Collaborative Group. N Engl J Med. 1995 Feb 9;332(6):345-50. doi: 10.1056/NEJM199502093320601. PMID 7823995
- [Result] Brochard L, Rauss A, Benito S, Conti G, Mancebo J, Rekik N, Gasparetto A, Lemaire F. Comparison of three methods of gradual withdrawal from ventilatory support during weaning from mechanical ventilation. Am J Respir Crit Care Med. 1994 Oct;150(4):896-903. doi: 10.1164/ajrccm.150.4.7921460.
- [Result] Esteban A, Alia I, Gordo F, Fernandez R, Solsona JF, Vallverdu I, Macias S, Allegue JM, Blanco J, Carriedo D, Leon M, de la Cal MA, Taboada F, Gonzalez de Velasco J, Palazon E, Carrizosa F, Tomas R, Suarez J, Goldwasser RS. Extubation outcome after spontaneous breathing trials with T-tube or pressure support ventilation. The Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):459-65. doi: 10.1164/ajrccm.156.2.9610109. PMID 9279224